CLINICAL TRIAL: NCT05404815
Title: Exposure to Plasticizers in the Neonatal Intensive Care Unit and Long- Term Neurodevelopmental and Pulmonary Toxicity
Brief Title: Exposure to Plasticisers in the Neonatal Intensive Care Unit
Acronym: PLASTIC-NICU
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Research Foundation Flanders (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: 20/23/022
Record Dates: First submitted 2022-05-13; First posted 2022-06-03 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2023-08

CONDITIONS: Preterm Birth; Premature Birth; Neurodevelopmental Disorders; Pulmonary Disease; Bronchopulmonary Dysplasia; Harm Reduction; Environmental Exposure; Development, Infant
Keywords: Plasticizers; Phthalates; Alternative Plasticizers; Respiratory development; Neurodevelopmental outcome; Preterm birth; Neonatal Intensive Care Unit; NICU
MeSH Terms: conditions — Premature Birth; Neurodevelopmental Disorders; Lung Diseases; Bronchopulmonary Dysplasia; Harm Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, hair, breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neonatal intensive care relies on indwelling plastic medical devices fundamental in respiratory support, intravenous catheterization, and nutrition. While being in a critical developmental period, constant exposure to these invasive medical devices puts premature neonates at risk of plasticizers' potential toxicity. Despite novel regulations and development of alternative plasticizers (AP), reference to guide manufacturers and an overview of the prevailing exposure levels to DEHP or alternatives in the neonatal intensive care unit (NICU) are still missing. The three main objectives of this project are: (1) to assess current exposure to plasticizers in the NICU, (2) to identify the sources of exposure and (3) to study the resultant long-term health risk in premature neonates. These objectives are addressed in three work packages (WP). In work package 1, in vivo exposure of premature neonates to phthalates and alternative plasticizers is assessed by determining their metabolites in biological matrices (urine and hair). Work package 2 explores ex vivo leaching characteristics of different plasticizers from medical devices used in the NICU. Finally, Work package 3 studies the long-term neurocognitive and lung development in relation to plasticizer exposure in the NICU.

DETAILED DESCRIPTION:
RESEARCH HYPOTHESIS: Leaching of plasticizers (DEHP and APs) from indwelling medical devices used in the neonatal intensive care unit (NICU) may expose premature neonates to these chemicals and their metabolites. The resulting exposure may contribute to medical risks and to impaired (neurocognitive) development of the children after hospital discharge.

This project aims to explore scalp hair and urine as a diagnostic tool for exposure to plasticizers in the extremely vulnerable population of premature neonates. The use of scalp hair to detect past exposure is by itself a novel approach and is expected to provide fresh insights into the role of plasticizers in post NICU morbidity. Within this project, we intend to address the following goals to be pursued:

Objective 1. Exploring the use of a non-invasive matrix (scalp hair) to determine past exposure to plasticizers in neonates. By measuring the levels of DEHP and AP metabolites A/ soon after birth in urine and neonatal scalp hair to determine intra-uterine exposure and B/ during follow-up after NICU discharge in infant scalp hair to determine past exposure in NICU (3 months) and early life (12 months).

Objective 2. To study the extent of leaching of plasticizers from indwelling medical devices used in NICU, by A/ determining the ex vivo leaching from the devices in ambient conditions and taking into account acidity and lipid content with relevance for neonatal care and B/ quantifying levels of plasticizers and metabolites in neonatal urine, collected on daily basis upon NICU admission until discharge.

Objective 3. To study the contribution of exposure to plasticizers leaching from indwelling medical devices used in the NICU, to neurocognitive and pulmonary development during the first year of life.

Importance and impact: NICU saves many lives of premature babies, but the long-term consequences of NICU may jeopardize the quality of life. Hence, finding strategies to prevent or attenuate this legacy is crucial. The completion of this project will lead to a comprehensive characterization of the potential health effects arising from leaching of plasticizers currently used in medical devices in NICU.

The study will be carried out in the NICU of the Antwerp University Hospital (UZA), a 28-beds ICU serving as a tertiary reference centre. We will include neonates with a gestational age under 31 weeks and/or birth weight under 1500 grams. We focus on this group of extreme premature neonates, because of their high and prolonged exposure. Board certified neonatologists will prospectively follow up the neonates. All are exposed to a variable number (range 1-6) of a diversity of indwelling medical devices, leading to a variable degree of exposure in the individual neonate. Term born neonates with age, gender and socio-economic status (not admitted to the NICU, n=100) comparable with those of the patients will be recruited as a control group for non-NICU exposure. The study protocol and informed consent forms have already been approved by the UZA Ethical Committee (Ref. 2003022).

ELIGIBILITY:
Inclusion Criteria:

* Preterm NICU neonates: Gestational Age < 31 weeks and/or birth weight < 1500 gram
* Healthy controls: term neonates

Exclusion Criteria:

* Major congenital abnormalities

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be carried out in the NICU of the Antwerp University Hospital (UZA), a 28-beds ICU serving as a tertiary reference centre. We will include neonates with a gestational age under 31 weeks and/or birth weight under 1500 grams. We focus on this group of extreme premature neonates, because of their high and prolonged exposure. Board certified neonatologists will prospectively follow up the neonates. All are exposed to a variable number (range 1-6) of a diversity of indwelling medical devices, leading to a variable degree of exposure in the individual neonate. Term born neonates with age, gender and socio-economic status (not admitted to the NICU, n=100) comparable with those of the patients will be recruited as a control group for non-NICU exposure.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Level and sources of NICU exposure to phthalates and alternative plasticizers, measured by liquid chromatography coupled to tandem mass spectrometry in urine samples. | Starting at day 1 postnatal, we collect weekly urine samples, until term age (40 weeks post-menstrual age) or NICU discharge (whatever comes first, up to 120 days postnatally).
  Urine samples are analysed for phthalate and alternative plasticizers' metabolites by liquid chromatography coupled to tandem mass spectrometry at the Antwerp Toxicological Centre. Results will be described as ng/mL.
Level and sources of NICU exposure to phthalates and alternative plasticizers, measured by liquid chromatography coupled to tandem mass spectrometry in hair samples. | Scalp hair samples are being collected at term age (37-40 weeks post menstrual age).
  Hair samples are analysed for phthalate and alternative plasticizers' metabolites by liquid chromatography coupled to tandem mass spectrometry at the Antwerp Toxicological Centre. Results will be described as ng/mg.
Perinatal Morbidity | NICU Discharge (or death, assessed up to 40 weeks post menstrual age)
  Prospective data collection
Perinatal Survival | NICU Discharge (or death, assessed up to 40 weeks post menstrual age)
  Prospective data collection
Respiratory development - 3 months | 3 months corrected for gestational age
  Respiratory questionnaire
Respiratory development - 12 months | 12 months corrected for gestational age
  Respiratory questionnaire
Neurodevelopmental outcome - 3 months | 3 months corrected for gestational age
  Bayley Scales of Infant and Toddler Development (BSID III) - Mean score 100 points, standard deviation 15 points. Higher score corresponds to better outcome
Neurodevelopmental outcome - 12 months | 12 months corrected for gestational age
  Bayley Scales of Infant and Toddler Development (BSID III) - Mean score 100 points, standard deviation 15 points. Higher score corresponds to better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Jorens, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital - Neonatal Intensive Care Unit, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lucas Panneel, Govindan Malarvannan, Philippe G. Jorens, Adrian Covaci & Antonius Mulder (2021) Plasticizers in the neonatal intensive care unit: A review on exposure sources and health hazards, Critical Reviews in Environmental Science and Technology, DOI: 10.1080/10643389.2021.1970455
- [Result] Panneel L, Cleys P, Breugelmans C, Christia C, Malarvannan G, Poma G, Jorens PG, Mulder A, Covaci A. Neonatal exposure to phthalate and alternative plasticizers via parenteral nutrition. Int J Pharm. 2023 Jan 25;631:122472. doi: 10.1016/j.ijpharm.2022.122472. Epub 2022 Dec 13. PMID 36526146
- [Result] Cleys P, Panneel L, Bombeke J, Dumitrascu C, Malarvannan G, Poma G, Mulder A, Jorens PG, Covaci A. Hair as an alternative matrix to assess exposure of premature neonates to phthalate and alternative plasticizers in the neonatal intensive care unit. Environ Res. 2023 Nov 1;236(Pt 2):116712. doi: 10.1016/j.envres.2023.116712. Epub 2023 Jul 22. PMID 37482128
- [Result] Vercauteren M, Panneel L, Jorens PG, Covaci A, Cleys P, Mulder A, Janssen CR, Asselman J. An Ex Vivo Study Examining Migration of Microplastics from an Infused Neonatal Parenteral Nutrition Circuit. Environ Health Perspect. 2024 Mar;132(3):37703. doi: 10.1289/EHP13491. Epub 2024 Mar 20. No abstract available. PMID 38506503
- [Result] Panneel L, Cleys P, Poma G, Ait Bamai Y, Jorens PG, Covaci A, Mulder A. Ongoing exposure to endocrine disrupting phthalates and alternative plasticizers in neonatal intensive care unit patients. Environ Int. 2024 Apr;186:108605. doi: 10.1016/j.envint.2024.108605. Epub 2024 Mar 28. PMID 38569425